CLINICAL TRIAL: NCT06280352
Title: Prospective Randomized Controlled Trial of Functionally Aligned Robotically Assisted Total Knee Arthroplasty vs Patient Specific Custom Made Total Knee Arthroplasty
Brief Title: Robotic Assisted vs Custom Made Total Knee Arthroplasty
Acronym: Knieathlon
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Austrian Workers Compensation Board Styria (Other)
Responsible Party: Principal Investigator, Antonio Klasan, Assistant Professor, MD, PhD, EMBA, Austrian Workers Compensation Board Styria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AUVA_Knieathlon_2024
Record Dates: First submitted 2024-02-05; First posted 2024-02-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Custom made Total Knee Arthroplasty (Experimental): Implant used is a patient specific custom made total knee Origin (Symbios, Symbios Orthopédie SA, Avenue des Sciences 1, 1400 Yverdon-les-Bains, Switzerland)
  Interventions: Device: Custom made Total Knee Arthroplasty
- Functionally aligned robotically assisted total knee arthroplasty (Active Comparator): Total Knee Implant Triathlon (Stryker, Kalamazoo, Michigan, U.S.) implanted using MAKO Rio Robotic Arm (Stryker)
  Interventions: Device: Functionally aligned robotically assisted total knee arthroplasty

INTERVENTIONS:
Device: Custom made Total Knee Arthroplasty — Total knee replacement, patient specific custom made total knee Origin (Symbios, Symbios Orthopédie SA, Avenue des Sciences 1, 1400 Yverdon-les-Bains, Switzerland)
  Arms: Custom made Total Knee Arthroplasty
Device: Functionally aligned robotically assisted total knee arthroplasty — Total knee replacement, Total Knee Implant Triathlon (Stryker, Kalamazoo, Michigan, U.S.) implanted using MAKO Rio Robotic Arm (Stryker), using functional alignment strategy
  Arms: Functionally aligned robotically assisted total knee arthroplasty

SUMMARY:
The goal of this clinical trial is to compare Robotic Assisted, functionally aligned vs Custom Made Total Knee Arthroplasty in patients with knee osteoarthritis. The main questions it aims to answer are:

* Which implant/philosophy yields better clinical outcomes?
* Which implant/philosophy yields better satisfaction?
* Which system is more OR efficient? Participants will be followed for 2 years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* - The patient is a male or non-pregnant female between the ages of 40 and 90 years
* The patient requires a primary total knee replacement
* Patient is deemed appropriate for a cruciate retaining knee replacement
* The patient has a primary diagnosis of osteoarthritis (OA)
* The patient has intact collateral ligaments
* The patient is able to undergo CT scanning of the affected limb
* The patient has signed the study specific, ethics-approved, informed consent document
* The patient is willing and able to comply with the specified pre-operative and post-operative clinical and radiographic evaluations

Exclusion Criteria:

* - The patient has a history of total, unicompartmental reconstruction or fusion of the affected joint
* Patient has had a previous osteotomy around the knee
* The patient is morbidly obese (BMI > 41)
* The patient has a deformity which will require the use of stems, wedges or augments
* The patient has a varus deformity ≥ 15°
* The patient has a valgus deformity >3°
* The patient has a neuromuscular or neurosensory deficiency, which would limit the ability to assess the performance of the device
* The patient is unable to speak German
* The patient is pregnant

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Clinical Outcome using the Forgotten Joint Score | 6 weeks, 3 months, 6 months, 12 months, 24 months
  Scale 0-100, higher score means better outcome

SECONDARY OUTCOMES:
Clinical outcomes using the Kujala anterior knee pain Score | preoperatively, 6 weeks, 3 months, 6 months, 12 months, 24 months
  Scale 0-100, higher score means better outcome
Patient satisfaction | preoperatively, 6 weeks, 3 months, 6 months, 12 months, 24 months
  Question "Are you satisfied with the outcome of your operation" using a Likert scale with 5 points: 1- very dissatisfied, 2-dissatisfied, 3 - neither satisfied nor dissatisfied, 4 - satisfied, 5 - very satisfied
Visual analog pain (VAS) scale | preoperatively, 6 weeks, 3 months, 6 months, 12 months, 24 months
  Scale 0-10, higher score means better outcome
Surgical and total theatre time | Perioperative phase
Opioid use | Intraoperative stay
  Total dosage of opioids, registered in Austria for pain management after knee replacement, administered to the patient during in-hospital stay: Hydromorphon, Tramadol, Oxycodone/Naloxon as well as number of ampules of Piritramid
Number of physiotherapy sessions | Intraoperative stay
Range of motion measurements (in degrees) | preoperatively, 6 weeks, 3 months, 6 months, 12 months, 24 months
  Measurement using a manual goniometer.
Radiographic data including radiolucent lines | preoperatively, 6 weeks, 3 months, 6 months, 12 months, 24 months
  Incidence of radiolucent lines >1 mm, with zones defined according to the New Knee Society Classification
Revision rate | Minimum 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - AUVA UKH Steiermark Standort Graz, Graz, Styria
  - AUVA UKH Steiermark Standort Kalwang, Kalwang, Styria

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT06280352/Prot_SAP_000.pdf